CLINICAL TRIAL: NCT03667976
Title: South Asian Women Together in a Health Initiative (SATHI): A Pilot Randomized Controlled Trial
Brief Title: South Asian Women Together in a Health Initiative: A Pilot RCT
Acronym: SATHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Abida Ramzan Dhukai, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35823
Record Dates: First submitted 2018-07-25; First posted 2018-09-12 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Women's Health
Keywords: cardiovascular disease; South Asian; physical activity; peer support; pedometer
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: A pragmatic two-arm parallel 12-week pilot randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The investigator will (a) screen, determine eligibility, and obtain consent from eligible peers, (b) schedule and deliver the peer training session, (c) provide support and answer questions of peers as required, (d) assist in the organization of peer meetings and discussions as required, and (e) will pair participants with the appropriate peer based on having children (peer-participant dyad) via telephone.
  The outcome assessor (research assistant) will be blinded. Study participants will be assigned a unique study identification (ID) number and will use this study ID number when they electronically submit step counts to the research assistant at weeks 6 and 12. Intervention group participants will additionally submit step counts weekly until study completion. All other outcome data will be collected by the research assistant at the 12-weeks post-intervention follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): All participants in the control group will receive a study pedometer and a physical activity logbook. Participants will also receive the Canadian Society of Exercise Physiology/ParticipACTION physical activity guidelines for adults ages 18 to 64.
- Intervention Group (Experimental): All participants in the intervention group will receive a study pedometer and a physical activity logbook. Participants will also receive the South Asian women Together in a Health Initiative (SATHI) intervention which consists of a gender and culturally specific South Asian physical activity education booklet and video and 2) a matched peer. Peers will encourage physical activity and provide motivation and suggestions for incorporating physical activity into daily life of a South Asian woman based on Bandura's Self-Efficacy construct. Peer contact will occur via telephone, text/email messaging or in person at least once weekly and more often as determined by participants.
  Interventions: Behavioral: SATHI

INTERVENTIONS:
Behavioral: SATHI — see above
  Arms: Intervention Group

SUMMARY:
The overall goal of this pilot study is to assess the feasibility, acceptability and potential effects of a culturally tailored 12-week peer-based physical activity intervention compared with a control group, among young sedentary Canadian South Asian women. Specific objectives are: 1) To determine the feasibility (recruitment, retention, engagement, and acceptability) of implementing the SATHI intervention, and 2) To determine the effect of the SATHI intervention on physical activity, anthropometric risk (waist circumference, waist-hip ratio, and body mass index), and self-efficacy.

This is an innovative, gender-specific and culturally tailored primary prevention intervention for South Asian women who are at increased risk of cardiovascular disease. Information obtained from this pilot trial will inform a larger multi-centred trial and will also help inform health care providers and researchers about novel means of researching, educating and engaging South Asians in healthy lifestyle behaviours relevant to their daily lives.

DETAILED DESCRIPTION:
Background. Canadian South Asian women have high rates of cardiovascular disease morbidity and mortality and the lowest rates of physical activity in Canada, which increases risk for type II diabetes mellitus, hypertension, obesity and cardiovascular disease.

The overall goal of this pilot randomized controlled trial is to assess the feasibility and acceptability of a culturally tailored 12-week peer-based physical activity intervention, among 48 sedentary Canadian South Asian women, ages 24 to 39, in the Greater Toronto Area. Specific objectives are to determine: 1) The feasibility (recruitment, retention, engagement, and acceptability) of implementing the South Asian women Together in a Health Initiative (SATHI) intervention, and 2) The effect of SATHI on physical activity (step count, moderate/vigorous physical activity, weight/resistance training), anthropometric risk (waist circumference, waist-to-hip ratio, body mass index), and self-efficacy (Physical Activity Appraisal Inventory).

Sample and Setting. Participants will include: 1) Canadian South Asian women, 2) aged 24 to 39 years, 3) sedentary, 4) without unstable medical or chronic conditions, and 5) residents of the Greater Toronto Area. All participants will be screened for safety using the Physical Activity Readiness Questionnaire-Plus screening tool. Peers will be: 1) Canadian South Asian women, 2) aged 24 and 39 years, and 3) who self-report achieving at least 30 minutes continuous moderate to vigorous physical activity five days per week. This trial will be conducted at community centres in the Greater Toronto Area.

Research Design. A pragmatic two-arm parallel 12-week pilot randomized controlled trial.

Recruitment. South Asian community centres will be used for participant and peer recruitment, data collection and intervention follow-up. Other strategies for participant and peer recruitment will include flyers distributed at the Punjabi Community Health Services, the multiservice centres at Peel Public Health, religious festivals, local mosques, temples, and gurudwaras, churches, South Asian restaurants, and grocery and clothing stores within the Greater Toronto Area. Popular female South Asian online personalities will also promote the study on social media.

Procedures. Upon completion of participant and peer recruitment, consent and collection of baseline demographic, anthropometric, and self-efficacy for exercise data, participants will be randomly allocated to either a control or intervention group, using block sizes of 4 and 8. All participants will receive a study pedometer, instructions on its use, and a physical activity logbook in which they will document daily step counts and physical activity. Control Group. Participants allocated to the control group will receive the Canadian Society of Exercise Physiology/ParticipACTION physical activity guidelines for adults ages 18 to 64. Intervention Group. Participants allocated to the intervention group will receive the: 1) South Asian physical activity education which includes a culturally specific physical activity education booklet and video and 2) peer support. Peers will encourage physical activity and provide motivation and suggestions for incorporating physical activity into daily life of a South Asian woman using Bandura's Self-Efficacy construct. Peer contact will occur via telephone/text/email messaging or in person at least once a week and more often as determined by participants. All peers will receive 4-hours of training and will be matched to participants based on presence of child(ren). Peers will not provide medical advice and will document all participant-peer interactions on a log sheet that will be submitted to the trial investigator.

Outcomes. Participants in control and intervention groups will submit baseline step counts. After randomization, intervention group participants will submit weekly step counts to the research assistant. All other outcome data will be collected at 12-weeks. Primary Outcomes. Participant and peer recruitment, retention, engagement, and acceptability rates for the SATHI intervention. Secondary Outcomes. Physical activity (step count, physical activity logbook), anthropometric measures (waist circumference, waist-to-hip ratio, body mass index) and self-efficacy (Physical Activity Appraisal Inventory).

Data Analysis. All statistical analysis will be completed using SPSS Statistics v.24. Descriptive statistics will be conducted to analyze baseline outcome measures. Paired t-tests will be used to assess between-group mean differences. Mean change scores (T2-T1) for both control and intervention groups will be calculated for within group differences. Since this is a feasibility trial, a p-value will be set at p<0.10.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Canadian South Asian women with ethnic roots from Indian, Pakistan, Bangladesh, Sri Lanka and Nepal
* 24 to 39 years of age
* self-report achieving less than 30 minutes of continuous moderate to vigorous physical activity on three days per week
* able to understand written and spoken English
* have access to a password protected computer, tablet or smartphone with a valid email address and telephone number
* a resident of the Greater Toronto Area for the duration of the study,
* answer "yes" to all seven questions of the Physical Activity Readiness Questionnaire-Plus (a physical activity safety screening tool).

Peers:

* Canadian South Asian women with ethnic roots from Indian, Pakistan, Bangladesh, Sri Lanka and Nepal
* 24 to 39 years of age
* self-report achieving at least 30 minutes continuous moderate to vigorous physical activity five days per week
* able to understand written and spoken English
* have access to a computer, tablet or smartphone with a valid email address and telephone number
* a resident of the Greater Toronto Area for the duration of the study.

Exclusion Criteria:

* attend a gym or physical activity classes for 30 minutes at least three times per week, or have a personal trainer
* participate in any prescribed or self-initiated program for weight loss
* have any known severe or chronic medical condition(s) that would prevent them from participating in the trial (e.g. uncontrolled diabetes mellitus defined as HbA1c ≥ 6.5%, uncontrolled hypertension defined as systolic blood pressure ≥130mmHg or diastolic blood pressure ≥80mmHg, unstable angina, symptomatic peripheral vascular disease [PVD], untreated depression, active treatment for depression with current adjustment of medications, cancer, chronic respiratory conditions such as severe asthma as defined as inability to control asthma despite the use of high dose treatment with inhaled corticosteroids, long-acting inhaled beta 2 agonists, montelukast, and/or theophylline, oral corticosteroid treatment for at least six months per year, or control is lost when treatment is decreased, or pulmonary fibrosis
* physical limitations preventing participation in study (e.g. blindness, deaf, wheelchair users)
* pregnant or lactating/breastfeeding women, or planning on becoming pregnant over the course of the study
* a family member/ friend of another SATHI participant

Ages: 24 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must self-identify as a woman.
Enrollment: 48 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Recruitment and Screening | Through study completion, an average of 6 months
  Number of participants and peers agreeing to participate compared to total screened
Recruitment and Participation | Through study completion, an average of 12 weeks
  Reasons for participant and peer non-participation
Recruitment Strategies | Through study completion, an average of 12 weeks
  Strategies for recruiting participants and peers
Retention Rates | Through study completion, an average of 12 weeks
  Participant and peer attrition
Retention Reasons | Through study completion, an average of 12 weeks
  Reasons for participant and peer attrition
Engagement in Physical Activity | Through study completion, an average of 12 weeks
  Number of participants who complete 60 minutes of physical activity daily
Engagement with Video | Through study completion, an average of 12 weeks
  Number of participants who watch the video
Engagement with Booklet | Through study completion, an average of 12 weeks
  Number of participants who read South Asian physical activity booklet
Engagement in Study | Through study completion, an average of 12 weeks
  Number of participants who complete the physical activity logbook daily and upload step count data every week
Engagement with Peer | Through study completion, an average of 12 weeks
  Participants who interact with peer at agreed upon intervals
Engagement of Peer | Through study completion, an average of 12 weeks
  Number of peers completing peer volunteer activity logs
Acceptability with Video | Through study completion, an average of 12 weeks
  Participant satisfaction with video
Acceptability with Peer | Through study completion, an average of 12 weeks
  Participant satisfaction with peer support
Acceptability Barriers Experienced | Through study completion, an average of 12 weeks
  Barriers to participant and peer participation
Acceptability of Orientation and Training | Through study completion, an average of 12 weeks
  Peer satisfaction with the orientation session and training manual
Acceptability and Physical Activity Strategies | Through study completion, an average of 12 weeks
  Commonly used strategies by participants to incorporate physical activity

SECONDARY OUTCOMES:
Physical Activity Step Count | At baseline and at study completion, an average of 12 weeks
  Step count
Physical Activity Logbook | At baseline and at study completion, an average of 12 weeks
  Physical activity logbook entries
Anthropometric Measures Waist Circumference | At baseline and at study completion, an average of 12 weeks
  Waist circumference
Anthropometric Measures Waist to Hip Ratio | At baseline and at study completion, an average of 12 weeks
  Waist-to-hip ratio
Anthropometric Measures BMI | At baseline and at study completion, an average of 12 weeks
  Body mass index
Self-efficacy for exercise | At baseline and at study completion, an average of 12 weeks
  Physical Activity Appraisal Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Abida R Dhukai, NP-A,PhD(c), Principal Investigator — University of Toronto
Locations (1):
- Peel Public Health, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data will be completely confidential and will not be shared with other researchers.